CLINICAL TRIAL: NCT01372423
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Multi-Site Study to Evaluate the Clinical Equivalence of Lubiprostone 24 Mcg Capsules (Anchen Pharmaceuticals, Inc.) With AMITIZA® (Lubiprostone) 24 Mcg Capsules (Sucampo Pharmaceuticals, Inc.) in the Treatment of Chronic Idiopathic Constipation
Brief Title: Evaluation of Clinical Equivalence Between Two Lubiprostone Products
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anchen Pharmaceuticals, Inc (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS-01-2011; 71060001 (Other: Novum Pharmaceutical Research Services)
Record Dates: First submitted 2011-06-10; First posted 2011-06-14 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Idiopathic Constipation
MeSH Terms: interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- AMITIZA (Active Comparator): Manufactured by Sucampo Pharmaceuticals (24 mcg administered for 7 days)
  Interventions: Drug: Lubiprostone
- Placebo (Placebo Comparator): Manufactured by Anchen Pharmaceuticals (24 mcg administered for 7 days)
  Interventions: Drug: Placebo
- Lubiprostone (Experimental): Manufactured by Anchen Pharmaceuticals (24 mcg administered for 7 days)
  Interventions: Drug: Lubiprostone

INTERVENTIONS:
Drug: Lubiprostone — 24 mcg capsules
  Arms: AMITIZA; Lubiprostone
Drug: Placebo — 24 mcg capsules
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the clinical equivalence and safety of the Test formulation of lubiprostone 24 mcg capsules compared to the marketed formulation AMITIZA® (lubiprostone) 24 mcg capsules (Sucampo Pharmaceuticals, Inc.) in patients with confirmed chronic idiopathic constipation.

ELIGIBILITY:
Main Inclusion Criteria:

1. 1. Male or non-pregnant females aged 18 and older with a clinical diagnosis of chronic idiopathic constipation defined as, on average, < 3 spontaneous bowel movements (SBMs) per week for the past 6 months and confirmed by daily diary during the 14 day baseline lead-in period. An SBM is defined as any bowel movement that did not occur within 24 hours after rescue medication use.
2. Have 1 or more of the following symptoms related to bowel movements for at least 6 months before the baseline visit and confirmed by daily diary during the 14 Day baseline period:

   * very hard (little balls) and/or hard stools for at least 25 percent of the bowel movements
   * sensation of incomplete evacuation following at least 25 percent of the bowel movements
   * straining at defecation at least a quarter of the time
3. Women of child-bearing potential must have a negative pregnancy test prior to beginning therapy and agree to use effective contraceptive methods during the study.
4. For patients aged < 50 years, documentation of the results of either a flexible sigmoidoscopy or colonoscopy performed within the 5 years prior to dosing, showing no mechanical bowel obstruction or organic disorders of the large Bowel.
5. For patients aged >/= 50 years, documentation of the results of either a barium enema with flexible sigmoidoscopy or colonoscopy performed within 1 year prior to dosing, showing no mechanical bowel obstruction or organic disorders of the large bowel.

Main Exclusion Criteria:

1. Females who are Pregnant, breast feeding, or planning a pregnancy.
2. Patients of any age with evidence of weight loss, anemia, or rectal bleeding AND without documentation of the results of either a flexible sigmoidoscopy or colonoscopy performed during the 6 months prior to dosing.
3. Patients that have documented mechanical bowel obstruction (e.g., bowel obstruction due to tumor, hernia), megacolon/megarectum, or diagnosis of pseudo-obstruction.
4. Any known or suspected organic disorders of the large or small bowel (e.g., inflammatory bowel disease, ulcerative colitis, Crohn's Disease) or constipation secondary to a documented cause (e.g., surgery, bowel resection)or acute hernia.
5. History of bowel resection.
6. Patients who are regularly using medications know to cause constipation (narcotics, calcium channel blockers, tricyclic antidepressants).
7. Hospitalized for any gastrointestinal or abdominal surgical procedure during the 3 months prior to dosing.
8. Clinically significant cardiovascular, liver, lung, neurologic, renal or psychiatric disorder, or clinically significant laboratory abnormalities.
9. Use of a systemic antibiotic within 4 weeks prior to the Screening Visit.
10. Participation in a study with any investigational medication within the past 30 days of screening for this study or previous participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Primary Analysis | Day 8
  Clinical equivalence of the Test and Reference treatments and the superiority of each active treatment over the Placebo in the change from baseline in mean number of SBM's during the 7 day randomization period of the study.

SECONDARY OUTCOMES:
Safety Analysis | Day 8
  The frequency and severity of adverse events across treatment groups will be analyzed.

CONTACTS AND LOCATIONS:
Locations (79):
- United States (79):
  - Novum Investigator Site, Dothan, Alabama
  - Novum Investigator Site, Huntsville, Alabama
  - Novum Investigator Site, Mobile, Alabama
  - Novum Investigator Site, Chandler, Arizona
  - Novum Investigator Site, Gilbert, Arizona
  - Novum Investigator Site, Mesa, Arizona
  - Novum Investigator Site, Phoenix, Arizona
  - Novum Investigator Site, Phoeniz, Arizona
  - Novum Investigator Site, Hot Springs, Arkansas
  - Novum Investigator Site, Little Rock, Arkansas
  - Novum Investigator Site, Mountain Home, Arkansas
  - Novum Investigator Site, Sherwood, Arkansas
  - Novum Investigator Site, Buena Park, California
  - Novum Investigator Site, Fresno, California
  - Novum Investigator Site, Garden Grove, California
  - Novum Investigator Site, La Palma, California
  - Novum Investigator Site, Long Beach, California
  - Novum Investigator Site, Sacremento, California
  - Novum Investigator Site, San Diego, California
  - Novum Invesitgator Site, San Ramon, California
  - Novum Investigator Site, Santa Ana, California
  - Novum Investigator Site, Westlake Village, California
  - Novum Investigator Site, Denver, Colorado
  - Novum Investigator Site, Wheat Ridge, Colorado
  - Novum Investigator Site, Adventura, Florida
  - Novum Investigator Site, Boyton Beach, Florida
  - Novum Investigator Site, Bradenton, Florida
  - Novum Investigator Site, Brookville, Florida
  - Novum Investigator Site, Clearwater, Florida
  - Novum Investigator Site, Deerfield Beach, Florida
  - Novum Investigator Site, Jupiter, Florida
  - Novum Investigator Site, Maimi, Florida
  - Novum Investigator Site, Miami, Florida
  - Novum Investigator Site, Niceville, Florida
  - Novum Investigator Site, Ormond Beach, Florida
  - Novum Investigator Site, Panama City, Florida
  - Novum Investigator Site, Port Orange, Florida
  - Novum Investigator Site, St. Petersburg, Florida
  - Novum Investigator Site, Tampa, Florida
  - Novum Investigator Site, West Palm Beach, Florida
  - Novum Investigator Site, Decauter, Georgia
  - Novum Investigator Site, Sandy Springs, Georgia
  - Novum Investigator Site, Stockbridge, Georgia
  - Novum Investigator Site, Lewiston, Idaho
  - Novum Investigator Site, Rockford, Illinois
  - Novum Investigator Site, Evansville, Indiana
  - Novum Investigator Site, Lexington, Kentucky
  - Novum Investigator Site, Shreveport, Louisiana
  - Novum Invesitgator Site, Hollywood, Maryland
  - Novum Investigator Site, Jackson, Mississippi
  - Novum Investigator Site, Mexico, Missouri
  - Novum Investigator Site, Washington, Missouri
  - Novum Investigator Site, Billings, Montana
  - Novum Investigator Site, Lincoln, Nebraska
  - Novum Investigator Site, Henderson, Nevada
  - Novum Investigator Site, Marlton, New Jersey
  - Novum Investigator Site, Newport News, New Jersey
  - Novum Investigator Site, Poughkeepsie, New York
  - Novum Investigator Site, Cary, North Carolina
  - Novum Investigator Site, Charlotte, North Carolina
  - Novum Investigator Site, High Point, North Carolina
  - Novum Investigator Site, Raleigh, North Carolina
  - Novum Investigator Site, Salisbury, North Carolina
  - Novum Investigator Site, Wilmington, North Carolina
  - Novum Investigator Site, Winstom-Salem, North Carolina
  - Novum Investigator Site, Beavercreek, Ohio
  - Novum Investigator Site, Centerville, Ohio
  - Novum Investigator Site, Sylvania, Ohio
  - Novum Investigator Site, Columbia, South Carolina
  - Novum Investigator Site, Chattanooga, Tennessee
  - Novum Investigator Site, Germantown, Tennessee
  - Novum Investigator Site, Hermitage, Tennessee
  - Novum Investigator Site, Houston, Texas
  - Novum Investigator Site, Longview, Texas
  - Novum Investigator Site, San Antonio, Texas
  - Novum Investigator Site, Sugarland, Texas
  - Novum Investigator Site, Charlottesville, Virginia
  - Novum Investigator Site, Virginia Beach, Virginia
  - Novum Investigator Site, Mountain Lake, Washington